CLINICAL TRIAL: NCT03927911
Title: A Multicenter, Prospective, Active Controlled, Real World, Phase 4 Study of EXPAREL in Multimodal Regimens Compared With Standard of Care for Postsurgical Pain Management in Subjects Undergoing Lumbar Posterior Spine Surgeries (FUSION)
Brief Title: Phase 4 Study in Adult Subjects Undergoing Posterior Lumbar Spine Surgeries
Acronym: FUSION
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to protocol feasibility given the rapid evolution of medical practice for spinal procedure. Data from approximately 65 FUSION study subjects will be analyzed with the intent to create either a future study or registry for this patient population.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-413
Record Dates: First submitted 2019-04-19; First posted 2019-04-25 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain Management
MeSH Terms: interventions — Bupivacaine; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Open or mini-open surgical technique cohort (Active Comparator): Local infiltration Analgesia administered (with EXPAREL and bupivacaine HCl) in EXPAREL arm within cohort. EXPAREL arm to be compared to SOC arm within cohort
  Interventions: Drug: EXPAREL and Bupivacaine; Drug: Standard of Care
- Tubular or Percutaneous cohort (Minimally Invasive Cohort) (Active Comparator): Local infiltration Analgesia administered (with EXPAREL and bupivacaine HCl) in EXPAREL arm within cohort. EXPAREL arm to be compared to SOC arm within cohort
  Interventions: Drug: EXPAREL and Bupivacaine; Drug: Standard of Care
- Lumbar decompression without fusion (Outpatient Cohort) (Active Comparator): Local infiltration Analgesia administered (with EXPAREL and bupivacaine HCl) in EXPAREL arm within cohort. EXPAREL arm to be compared to SOC arm within cohort
  Interventions: Drug: EXPAREL and Bupivacaine; Drug: Standard of Care

INTERVENTIONS:
Drug: EXPAREL and Bupivacaine — Drug: EXPAREL and Bupivacaine HCl 0.5%
Drug: Standard of Care — Standard of Care

SUMMARY:
Primary Objective: The primary objective of this study is to compare postsurgical opioid consumption through 72 hours postsurgery in patients receiving local infiltration analgesia (LIA) with EXPAREL and bupivacaine HCl (EXPAREL group) with that of patients receiving standard of care (SOC) (control group) in adult subjects undergoing posterior lumbar spine surgeries where both groups are receiving a multimodal pain regimen.

Secondary Objectives: The secondary objectives of this study are to:

1. Compare safety and effectiveness outcomes following LIA with EXPAREL and bupivacaine hydrochloride (HCl) versus SOC in adult subjects undergoing posterior lumbar spine surgeries through 72 hours, including time to first opioid and opioid-related adverse events (ORAEs).
2. Compare health outcomes following LIA with EXPAREL and bupivacaine hydrochloride (HCl) versus SOC in adult subjects undergoing posterior lumbar spine surgeries, including discharge readiness, hospital (or other facility) length of stay (LOS), discharge disposition, hospital readmissions, and health service utilization.

DETAILED DESCRIPTION:
This is a Phase 4, multicenter, prospective, active-controlled, real world, study in approximately 225 adult subjects undergoing posterior lumbar spine surgery under general anesthesia.

Subjects will be screened within 30 days prior to surgery; screening on the day of surgery will be allowed but is discouraged. If a subject can only be screened on the day of surgery, the informed consent process must still be started at least 24 hours prior to the conduct of any screening procedures that are not considered SOC at the institution and such procedures may not be performed until written informed consent is provided. All screening procedures that are not SOC must be performed and documented within the 30-day time window (inclusive of the day of surgery for those subjects who can only be screened on the day of surgery) as described here.

During the screening visit, subjects will be assessed for any past or present medical conditions that in the opinion of the investigator would preclude them from study participation. After the ICF is signed, the following information will be recorded and procedures done: medical history, surgical history, medication history, the subject's opioid use history will be recorded to calculate mean daily mg oral morphine equivalent dosing (MED PO) in the last 30 days, demographic and background information, height, weight and body mass index (BMI), a urine pregnancy test for women of childbearing potential, and the subject's current adverse experiences (AEs), if any.

Subjects will be asked questions and/or be asked to fill forms as part of the following assessments: Brief Pain Inventory - short form (BPI-sf), 5-item Opioid Compliance Checklist (OCC), Hospital Anxiety and Depression Scale (HADS), Survey of Pain Attitudes (SOPA), Numeric Rating Scale (NRS) ti assess pain and Opioid Related Symptom Distress Scale (ORSDS).

Based on the planned surgical procedure, subjects will be placed in one of three cohorts:

* Cohort 1 - Open lumbar spinal fusion technique; ("open" cohort)
* Cohort 2 - Minimally invasive tubular and/or percutaneous pedicle screw insertion for lumbar decompression with or without fusion;("tubular/percutaneous without midline incision" cohort)
* Cohort 3 - Lumbar decompression surgery (LDS) without fusion (discectomy or laminectomy outpatient cohort)

The initial sample size in each study cohort (i.e., cohort 1, cohort 2 and cohort 3) is estimated at 75 subjects (50 subjects with EXPAREL and 25 subjects with Control group), for a total of 225 subjects in all three cohorts. Within each assigned cohort, subjects will be allocated in a 2:1 ratio to the EXPAREL (50 subjects) and Control group (25 subjects).

The following sequence will be followed for all cohorts: First, the subjects who meet eligibility criteria will be treated according to the institution's SOC. Their data will be collected prospectively. Next, at each investigational site, the administration of EXPAREL and bupivacaine HCl to the first 1 to 3 subjects in each cohort will be observed to ensure that the correct procedure for infiltration as described in the infiltration guide is being followed. If the infiltration was performed correctly, the subject will be included in the study. If the infiltration was performed incorrectly, the subject will continue in the study but will be removed from statistical analysis and will be replaced to ensure at least 50 evaluable EXPAREL patients are enrolled per cohort. If subjects are discontinued for other reasons, they will be replaced such that a total sample size of 75 fully evaluable subjects is obtained in each study cohort, with 50 in the EXPAREL group and 25 in the Control group.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old at the time of screening.
2. Primary surgical indication is related to spinal degenerative disease, including any of the following:

   1. Spinal stenosis
   2. Spondylolisthesis
   3. Radiculopathy/instability disc disorders
   4. Degenerative disc disease
3. Medically cleared for elective spine surgery.
4. Scheduled to undergo:

   1. Elective (i.e., not emergency)
   2. Lumbosacral (i.e., L1-S1)
   3. Posterior approach with posterior instrumentation
5. Cohort 1 - Open only:

   Open or mini-open surgical technique with:
   1. 1-level (i.e., spanning 2 vertebrae) or 2-level (i.e., spanning 3 contiguous vertebrae)
   2. Primary fusion or revision fusion
   3. Open or mini-open surgical technique
6. Cohort 2 - Tubular or percutaneous cohort only:

   1. 1-level (i.e., spanning 2 vertebrae) or 2-level (i.e., spanning 3 contiguous vertebrae)
   2. Primary fusion or revision fusion
   3. Tubular or percutaneous surgical technique
7. Cohort 3 - Lumbar decompression without fusion outpatient cohort only:

   1. Radiculopathy
   2. Spinal stenosis
8. Able to provide informed consent and adhere to all study assessments and visit schedule

Exclusion Criteria:

1. Serious spinal pathology determined by Investigator that might meaningfully affect postsurgical outcomes, including any of the following:

   1. Suspected cauda equina syndrome (e.g., bowel/bladder involvement)
   2. Infection
   3. Tumor
   4. Fracture
   5. Systemic inflammatory spondyloarthropathy
2. Contraindication to local anesthesia according to the clinical judgment of the Investigator and based on the EXPAREL label.
3. Patients who most likely will require patient-controlled analgesia (PCA) pumps in EXPAREL group.
4. Anterior surgical approaches, including any of the following:

   1. Anterior lumbar interbody fusion (ALIF)
   2. Oblique lumbar interbody fusion (OLIF)
   3. Anterior-posterior or 360º fusion
5. Lateral surgical approaches, including any of the following:

   1. Extreme lateral interbody fusion (XLIF)
   2. Direct lateral interbody fusion (DLIF)
6. High-dose presurgical opioid use:

   a) Mean daily intake greater than 100 mg mEq PO in the past 30 days
7. Known allergy, hypersensitivity, or contraindication to any of the following study medications:

   1. Bupivacaine
   2. EXPAREL
   3. Tylenol (acetaminophen)
   4. Robaxin
   5. 2 or more NSAIDs
   6. 2 or more gabapentinoids
   7. 2 or more rescue opioids (e.g., oxycodone, morphine, hydromorphone)
   8. 2 or more medications for postoperative nausea, vomiting, or pruritus (e.g., dexamethasone, ondansetron)
8. History of severely impaired renal or hepatic function.
9. Severe chronic pain that requires analgesic treatment, and in the opinion of the principal Investigator, is likely to meaningfully affect postsurgical outcomes.
10. Subjects that have implanted spinal cord stimulator or intrathecal drug pump.
11. Any neurologic or psychiatric disorder that might impact postsurgical pain or interfere with study assessments per Investigator discretion.
12. Malignancy in the last 2 years.
13. History of misuse, abuse, or dependence on opioid analgesics, other prescription drugs, illicit drugs, or alcohol as defined in DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition). Dependence or chronic opioid use will be defined as use of more than 30 morphine equivalents per day during the prior 90 days.
14. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
15. Body Mass Index < 17 kg/m2 or >44 kg/m2 at screening
16. Subjects receiving Worker's Compensation for disability or who are involved in other litigation related to the spine.
17. Planned concurrent surgical procedure.
18. Previous participation in an EXPAREL study.
19. Administration of any investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

In addition, the subject might be excluded from the study prior to study drug infiltration if one of the following criteria during the surgical procedure is met:

1. Unable to place planned surgical instrumentation
2. Poor fixation at the time of surgical instrumentation

In addition, the subject must be considered an early termination if one of the following criteria after the surgical procedure is met:

1. An incision size >20 cm
2. Autograft taken from a harvest site other than surgical site (i.e., iliac crest autograft)
3. Intraoperative complications likely to meaningfully affect postsurgical outcomes, including any of the following:

   1. Clinically significant and prolonged (i.e., >24 hours) neurologic deficit (e.g., foot drop)
   2. Dural tear or suspected dural tear requiring bed rest (exception: subject will be allowed if the dural tear is fixed as per SOC of the institution during surgery)
   3. Extensive bleeding (i.e., >1,000 mL blood loss)
   4. Symptomatic epidural hematoma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Nevins, DC, Study Director — Pacira Pharmaceuticals, Inc
Locations (12):
- United States (12):
  - Yale School of Medicine, New Haven, Connecticut
  - Marcus Neuroscience Institute, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - The Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Carolina NeuroSurgery & Spine Associates, P.A., Charlotte, North Carolina
  - M3-Emerging Medical Research, LLC, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Summit Spine Institute, Portland, Oregon
  - First Surgical Hospital, Bellaire, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subject might be excluded from the study prior to study drug infiltration if one of the following criteria during the surgical procedure is met:
  1. Unable to place planned surgical instrumentation
  2. Poor fixation at the time of surgical instrumentation
Groups:
- Cohort 1:Open or Mini-open Surgical Technique; Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort); Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort): Local infiltration Analgesia administered (with EXPAREL and bupivacaine HCl) in EXPAREL arm within cohort. EXPAREL arm to be compared to SOC arm within cohort
  EXPAREL and Bupivacaine: Drug: EXPAREL and Bupivacaine HCl 0.5%
  Standard of Care: Standard of Care
- Cohort 1 Control Group; Cohort 2 Control Group; Cohort 3 Control Group: Standard of Care
Period: Overall Study
Arm/Group | Cohort 1:Open or Mini-open Surgical Technique | Cohort 1 Control Group | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) | Cohort 2 Control Group | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) | Cohort 3 Control Group
Started | 0 | 17 | 0 | 3 | 13 | 32
Completed | 0 | 15 | 0 | 1 | 13 | 25
Not Completed | 0 | 2 | 0 | 2 | 0 | 7
Not completed — problems with eDiary | 0 | 1 | 0 | 1 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — not treated -study terminated by sponsor | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Surgery cancelled | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Trial was terminated, not all arms had participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1:Open or Mini-open Surgical Technique | Cohort 1 Control Group | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) | Cohort 2 Control Group | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) | Cohort 3 Control Group | Total
Number analyzed (Participants) | 0 | 17 | 0 | 3 | 13 | 32 | 65
Age, Continuous [Mean (Full Range); unit: years] |  | 60.94 [47 to 75] |  | 56 [53 to 60] | 52.38 [22 to 74] | 52.66 [21 to 72] | 55.495 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 0 | 0 | 9 | 11 | 28
  Male | 0 | 9 | 0 | 3 | 4 | 21 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 16 | 0 | 3 | 12 | 27 | 58
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0 | 0 | 0 | 0
  Asian |  | 0 |  | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0 | 0 | 0 | 0
  Black or African American |  | 1 |  | 0 | 0 | 1 | 2
  White |  | 15 |  | 3 | 12 | 29 | 59
  More than one race |  | 0 |  | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 1 |  | 0 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States |  | 17 |  | 3 | 13 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Post-surgical Opioid Consumption in mg MED PO (0-72 Hours)
Description: Post-surgical opioid consumption in mg MED PO from 0 hours (end of surgery) to 72 hours postsurgery
Time Frame: 0-72 hours
Population: Trial was terminated, not all arms had participants enrolled.
Measure: Mean (Standard Deviation); unit: MED, mg
Arm/Group | Cohort 1:Open or Mini-open Surgical Technique | Cohort 1 Control Group | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) | Cohort 2 Control Group | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) | Cohort 3 Control Group
Number analyzed (Participants) | 0 | 16 | 0 | 2 | 13 | 30
MED, mg |  | 90.7 (96.91) |  | 56.8 (5.30) | 51.6 (60.98) | 83.6 (109.84)

2. Secondary Outcome: Post-surgical Opioid Consumption in mg MED PO at 14 Days After Surgery
Description: Post-surgical opioid consumption in mg MED PO at 14 days after surgery
Time Frame: 0-14 days after surgery
Population: Trial was terminated, not all arms had participants enrolled.
Measure: Mean (Standard Deviation); unit: MED, mg
Arm/Group | Cohort 1:Open or Mini-open Surgical Technique | Cohort 1 Control Group | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) | Cohort 2 Control Group | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) | Cohort 3 Control Group
Number analyzed (Participants) | 0 | 16 | 0 | 2 | 13 | 30
MED, mg |  | 279 (330.66) |  | 330.8 (42.78) | 158.4 (242.71) | 187.7 (252.40)

3. Secondary Outcome: Time to First Opioid Rescue Through 72 Hours or Discharge.
Description: Time to first opioid rescue through 72 hours or discharge.
Time Frame: 0-72 hours
Population: Trial was terminated, not all arms had participants enrolled.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1:Open or Mini-open Surgical Technique | Cohort 1 Control Group | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) | Cohort 2 Control Group | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) | Cohort 3 Control Group
Number analyzed (Participants) | 0 | 16 | 0 | 2 | 13 | 30
hours |  | 0.82 [0.58 to 8.02] |  | 0.36 [0.03 to 0.68] | 3.07 [0.60 to 25.10] | 0.95 [0.83 to 1.52]

ADVERSE EVENTS:
Time Frame: AEs were collected from time of signing informed consent to Day 30 phone call.
Description: Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Groups:
- Cohort 1 Control Group: Standard of Care for open or mini-open surgical technique cohort
- Cohort 2 Control Group: Standard of Care for Tubular or Percutaneous Cohort (Minimally Invasive Cohort)
- Cohort 3 Control Group: Standard of Care for Limbar decompression without fusion (Outpatient Cohort)
Arm/Group | Cohort 1:Open or Mini-open Surgical Technique | Cohort 1 Control Group | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) | Cohort 2 Control Group | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) | Cohort 3 Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/16 | 0/0 | 0/2 | 0/13 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/16 | 0/0 | 0/2 | 1/13 | 1/30
Other Adverse Events (participants affected / at risk) | 0/0 | 6/16 | 0/0 | 0/2 | 8/13 | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1:Open or Mini-open Surgical Technique (N=0) | Cohort 1 Control Group (N=16) | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) (N=0) | Cohort 2 Control Group (N=2) | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) (N=13) | Cohort 3 Control Group (N=30)
Cauda equina syndrome (Nervous system disorders) | NA | NA | NA | NA | 1 (1) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | NA | NA | NA | NA | 0 (0) | 1 (1)
Spinal epidural haematoma (Nervous system disorders) | NA | NA | NA | NA | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1:Open or Mini-open Surgical Technique (N=0) | Cohort 1 Control Group (N=16) | Cohort 2: Tubular or Percutaneous (Minimally Invasive Cohort) (N=0) | Cohort 2 Control Group (N=2) | Cohort 3: Lumbar Decompression Without Fusion (Outpatient Cohort) (N=13) | Cohort 3 Control Group (N=30)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (9)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extradural Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purulent discharge (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stitch abcess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03927911/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03927911/SAP_001.pdf